CLINICAL TRIAL: NCT01816594
Title: NeoPHOEBE: Pi3k Inhibition in Her2 OverExpressing Breast cancEr: A Phase II, Randomized, Parallel Cohort, Two Stage, Double-blind, Placebo-controlled Study of Neoadjuvant Trastuzumab Versus Trastuzumab + BKM120 in Combination With Weekly Paclitaxel in HER2-positive, PIK3CA Wild-type and PIK3CA Mutant Primary Breast Cancer
Brief Title: NeoPHOEBE: Neoadjuvant Trastuzumab + BKM120 in Combination With Weekly Paclitaxel in HER2-positive Primary Breast Cancer
Acronym: NeoPHOEBE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Breast International Group (Other); GBG Forschungs GmbH (Other); SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBKM120F2203
Record Dates: First submitted 2013-03-14; First posted 2013-03-22 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: HER2-positive Newly Diagnosed, Primary Breast Cancer
Keywords: HER2; breast cancer; neoadjuvant; PI3K inhibitor; first line chemotherapy; trastuzumab; GBG; SOLTI; BIG
MeSH Terms: conditions — Breast Neoplasms | interventions — NVP-BKM120; Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BKM120 + Trastuzumab + paclitaxel (Experimental): BKM120 (oral, pan-class I PI3K inhibitor) in combination with trastuzumab and paclitaxel.
  Interventions: Drug: BKM120; Drug: Trastuzumab; Drug: Paclitaxel
- BKM120 PBO + Trastuzumab + paclitaxel (Placebo Comparator): BKM120 placebo in combination with trastuzumab and paclitaxel
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: BKM120 Placebo

INTERVENTIONS:
Drug: BKM120 — Neo-adjuvant BKM120 (oral pan-class I PI3K inhibitor, continuous daily dosing). BKM120 was administered orally 100 mg/day.
  Other Names: Buparsilib
  Arms: BKM120 + Trastuzumab + paclitaxel
Drug: Trastuzumab — Trastuzumab is a humanized monoclonal antibody directed against the extracellular juxtamembrane domain of the HER2 receptor. Administered 4mg/kg i.v. load followed by 2mg/kg i.v. weekly.
Drug: Paclitaxel — Paclitaxel is a cytotoxic agent with proven antitumor activity in a variety of solid tumors. The antitumor activity of paclitaxel is based on tubulin-binding and stabilization of non-functional microtubule bundles, thereby blocking normal mitotic spindle development and subsequent cell division. Administered weekly 80mg/m2 i.v.
Drug: BKM120 Placebo — Neoadjuvant BKM120 placebo Administered orally 100 mg/day.
  Arms: BKM120 PBO + Trastuzumab + paclitaxel

SUMMARY:
This randomized, parallel cohort, two stage, double-blind, placebo-controlled study evaluated the oral PI3K inhibitor BKM120 in combination with trastuzumab and paclitaxel in HER2-positive, PIK3CA wild-type and PIK3CA mutant primary breast cancer prior to surgery (neo-adjuvant setting).

DETAILED DESCRIPTION:
NeoPHOEBE evaluated the efficacy (as defined by pCR) of BKM120 (an oral PI3K inhibitor) in combination with trastuzumab and paclitaxel in a randomized, placebo-controlled, neo-adjuvant study in women diagnosed with primary breast cancer >1.5 cm (by US or MRI) with centrally confirmed HER2 overexpression or amplification, who have not previously undergone treatment for invasive breast cancer.

Prior to the initiation of paclitaxel, there was a 6-week "biologic window" with trastuzumab plus BKM120 or placebo only. The study was conducted separately in two cohorts (PIK3CA mutated and PI3K3CA wild-type) using a two-stage approach. Within each cohort patients were randomized into one of the following treatment arms:

Arm 1: BKM120 plus trastuzumab for 6 weeks followed by BKM120 and trastuzumab plus weekly paclitaxel for an additional 12 weeks.

Arm 2: BKM120 placebo plus trastuzumab for 6 weeks followed by BKM120 placebo plus trastuzumab plus weekly paclitaxel for an additional 12 weeks.

After completion of study treatment, patients were to have undergone definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient had provided a signed study ICF prior to any screening procedure
* Patient was a female ≥ 18 years of age
* Patient has an ECOG performance status of 0-1
* Patient has a unilateral (multifocal or multicentric disease allowed), histologically confirmed, newly diagnosed early breast cancer >2cm by clinical examination and/or >1.5 cm confirmed by ultrasound or by MRI
* Patient has tumor tissue available for central review of ER, HER2 and PI3K status with centrally confirmed HER2-positive disease and known PI3KCA mutation status
* Patient has adequate bone marrow, renal and liver function
* Patient is able to swallow and retain oral medication

Exclusion Criteria:

* Patient has received prior systemic treatment for currently diagnosed disease
* Patient has a known contraindications, hypersensitivity or intolerance to trastuzumab, paclitaxel or products containing cremophor
* Patient has bilateral breast cancer or metastatic disease or inflammatory breast cancer
* LVEF below 50% as determined by MUGA scan or ECHO
* Patient has active cardiac disease or a history of cardiac abnormalities as defined in the protocol
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120
* Patient is currently receiving warfarin or other coumarin derived anti-coagulants
* Patient is currently receiving chronic treatment with corticosteroids or another immunosuppressive agents (standard premedication for paclitaxel and local applications allowed)
* Patient is currently receiving treatment with drugs known to be strong inhibitors or inducers of CYP3A
* Patient has certain scores on an anxiety and depression mood questionnaires
* Pregnant or nursing (lactating) women or patients not willing to apply apply highly effective contraception as defined in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2015-02-18 (Actual); Study Completion 2015-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Salzburg, Austria
- Germany (2):
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Offenbach
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Loibl S, de la Pena L, Nekljudova V, Zardavas D, Michiels S, Denkert C, Rezai M, Bermejo B, Untch M, Lee SC, Turri S, Urban P, Kummel S, Steger G, Gombos A, Lux M, Piccart MJ, Von Minckwitz G, Baselga J, Loi S. Neoadjuvant buparlisib plus trastuzumab and paclitaxel for women with HER2+ primary breast cancer: A randomised, double-blind, placebo-controlled phase II trial (NeoPHOEBE). Eur J Cancer. 2017 Nov;85:133-145. doi: 10.1016/j.ejca.2017.08.020. Epub 2017 Sep 17. PMID 28923573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned: Minimum 128 patients (in case of early stopping of both cohorts), maximum: 220 patients (if both cohorts would have proceeded into stage 2), and 174 patients if one cohort would have stopped early.
Pre-assignment Details: Screened: 68 patients Randomized and analyzed (safety and efficacy): 50 patients
Groups:
- Trastuzumab + BKM120 + Paclitaxel: BKM120 (oral, pan-class I PI3K inhibitor) in combination with trastuzumab and paclitaxel.
- Trastuzumab + BKM120 PBO + Paclitaxel: BKM120 placebo in combination with trastuzumab and paclitaxel
Period: Overall Study
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Started | 25 | 25
Randomized to the wt Cohort | 21 (wt = PIK3CA wild-type) | 21 (wt = PIK3CA wild-type)
Randomized to the mt Cohort | 4 (mt = PIK3CA mutant) | 4 (mt = PIK3CA mutant)
Completed | 14 | 23
Not Completed | 11 | 2
Not completed — Local Progress | 0 | 2
Not completed — Adverse Event | 9 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients (N=50) were included in the intention-to-treat set and in the safety analysis set, since all patients started study treatment. Intent-to-treat set (ITT)/full analysis set (FAS) (pooled): The full analysis set comprised all patients to whom study treatment had been assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (11.5) | 51.3 (11.2) | 51.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/white | 21 | 24 | 45
  Asian/Oriental | 3 | 1 | 4
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response (pCR) Rate at the Time of Surgery - All Participants
Description: Rate of pCR (as defined by NSABP criteria - absence of invasive disease in the breast [ypT0]) is the number of of participants with pathological complete response (pCR) at the time of surgery. Participants were to be considered in pCR if there was no invasive cancer in the breast or only non-invasive in situ cancer in the breast specimen. NSABP guidelines do not take into account the histological nodal status to define the pCR.
Time Frame: After 6 weeks
Population: Intent-to-treat set (ITT)/full analysis set (FAS) (pooled): The full analysis set comprised all patients to whom study treatment had been assigned by randomization. Patients who were randomized but did not start study treatment were not replaced and were considered as treatment failures similarly to other patients with no pCR assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 32.0 [14.9 to 53.5] | 40.0 [21.1 to 61.3]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; All participantss; Test type: Superiority; p = 0.811, Fisher Exact; (one-sided)

2. Primary Outcome: Pathological Complete Response (pCR) Rate at the Time of Surgery - PIK3CA Wild Type (WT)
Description: as for outcome 1
Time Frame: After 6 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 21 | 21
Percentage of participants | 33.3 [14.6 to 57.0] | 42.9 [21.8 to 66.0]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; wild type cohort; Test type: Superiority; p = 0.830, Fisher Exact; (one-sided)

3. Primary Outcome: Pathological Complete Response (pCR) Rate at the Time of Surgery - PIK3CA Mutant (MT)
Description: as for outcome 1
Time Frame: After 6 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 4 | 4
Percentage of participants | 25.0 [0.6 to 80.6] | 25.0 [0.6 to 80.6]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; mutant cohort; Test type: Superiority; p = 0.786, Fisher Exact; (one-sided)

4. Secondary Outcome: Overall Objective Clinical Response Rate at the End of the Biologic Window (After Week 6) Compared to Baseline (Key Secondary) - All Participants
Description: Percentage of Overall objective clinical response rate = Complete Response + Partial Response rate, measured by US bidimentional ulltrasound (or MRI) and assessed by world health organization (WHO) criteria.
Time Frame: After week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 56.0 [34.9 to 75.6] | 44.0 [24.4 to 65.1]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; All participants; Test type: Superiority; p = 0.286, Fisher Exact; (one-sided)

5. Secondary Outcome: Overall Objective Clinical Response Rate at the End of the Biologic Window (After Week 6) Compared to Baseline (Key Secondary) - PIK3A Wild Type Participants
Description: as for outcome 4
Time Frame: After week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 21 | 21
Percentage of participants | 61.9 [38.4 to 81.9] | 42.9 [21.8 to 66.0]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; wild type cohort; Test type: Superiority; p = 0.177, Fisher Exact; (one-sided)

6. Secondary Outcome: Overall Objective Clinical Response Rate at the End of the Biologic Window (After Week 6) Compared to Baseline (Key Secondary) - PIK3A Mutant Participants
Description: as for outcome 4
Time Frame: After week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 4 | 4
Percentage of participants | 25.0 [0.6 to 80.6] | 50.0 [6.8 to 93.2]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; mutant cohort; Test type: Superiority; p = 0.929, Fisher Exact; (one-sided)

7. Secondary Outcome: Rate of Breast Conserving Surgery (Most Radical Surgery)
Description: Rate of patients with breast conserving surgery. Participants who did not have breast surgery were also considered as having breast conservation surgery (BCS)
Time Frame: 18 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 60.0 [38.7 to 78.9] | 68.0 [46.5 to 85.1]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; Test type: Superiority; p = 0.811, Fisher Exact; (one-sided)

8. Secondary Outcome: Percentage of Participants With No Invasive and Non-invasive (DCIS) Residuals in Breast and Lymph Nodes Per GBG Definition
Description: Rate of pCR defined as no invasive and non-invasive (DCIS) residuals in breast and lymph nodes (ypT0, ypN0 [GBG definition]). If patient had a sentinel node biopsy before treatment which was negative and no axilla dissection was performed after treatment completion, such patient was considered to be pN0 for both secondary pCR definitions. Surgical breast and axillary node resection specimens were evaluated for pathologic tumor response according to NSABP guidelines.
Time Frame: After Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 20.0 [6.8 to 40.7] | 28.0 [12.1 to 49.4]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; Test type: Superiority; p = 0.840, Fisher Exact; (one-sided)

9. Secondary Outcome: Percentage of Participants With No Invasive and Non-invasive (DCIS) Residuals in Breast and Lymph Nodes Per MD Anderson Definition
Description: Rate of pCR defined as no invasive residuals in breast and lymph nodes (ypT0/Tis, ypN0 [MD Anderson definition]). If a patient had a sentinel node biopsy before treatment which was negative and no axilla dissection was performed after treatment completion, such patient was considered to be pN0 for both secondary pCR definitions.
Time Frame: After Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 32.0 [14.9 to 53.5] | 36.0 [18.0 to 57.5]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; Test type: Superiority; p = 0.724, Fisher Exact; (one-sided)

10. Secondary Outcome: Overall Objective Response Rate (ORR) Prior to Surgery for All Participants
Description: Number of Overall objective response rate = Complete Response + Partial Response rate, measured by US bidimentional ulltrasound (or MRI) and assessed by world health organization (WHO) criteria. CR: Complete disappearance of all tumor signs in the breast as assessed by ultrasound or MRI. The response of the axillary nodes was not to be considered. PR: Reduction in the product of the two largest perpendicular diameters of the primary tumor size by 50% or more assessed by ultrasound or MRI. In patients with multifocal or multicentric disease, the lesion with the largest diameters should be chosen for follow-up. The response of the axillary nodes was not to be considered.
Time Frame: prior to surgery
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 56.0 [34.9 to 75.6] | 76.0 [54.9 to 90.6]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; All participants; Test type: Superiority; p = 0.964, Fisher Exact; (one-sided)

11. Secondary Outcome: Percentage of Participants With pCR Rates by Hormone Receptor Status - Positive Estrogen Receptor (ER+)
Description: pCR defined as no invasive and non-invasive (DCIS) residuals in breast and lymph nodes (ypT0, ypN0 [GBG definition]); pCR defined as no invasive residuals in breast and lymph nodes (ypT0/Tis, ypN0 [MD Anderson definition]). If participant had a sentinel node biopsy before treatment which was negative and no axilla dissection was performed after treatment completion, such participant was considered to be pN0 for both secondary pCR definitions.
Time Frame: After Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Trastuzumab + BKM120 + Paclitaxel ( ER+): BKM120 (oral, pan-class I PI3K inhibitor) in combination with trastuzumab and paclitaxel in positive estrogen receptor participants.
- Trastuzumab + BKM120 PBO + Paclitaxel (ER+): BKM120 placebo in combination with trastuzumab and paclitaxel in patients with positive estrogen receptor participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel ( ER+) | Trastuzumab + BKM120 PBO + Paclitaxel (ER+)
Number analyzed (Participants) | 16 | 15
Percentage of participants | 31.3 [11.0 to 58.7] | 26.7 [7.8 to 55.1]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel ( ER+) vs Trastuzumab + BKM120 PBO + Paclitaxel (ER+); For ER+ participants - pCR; Test type: Superiority; p = 0.546, Fisher Exact; (one-sided)

12. Secondary Outcome: Percentage of Participants With pCR Rates by Hormone Receptor Status Negative Estrogen Receptor (ER-)
Description: as for outcome 11
Time Frame: After Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Trastuzumab + BKM120 + Paclitaxel (ER-): BKM120 (oral, pan-class I PI3K inhibitor) in combination with trastuzumab and paclitaxel in negative estrogen receptor participants.
- Trastuzumab + BKM120 PBO + Paclitaxel (ER-): BKM120 placebo in combination with trastuzumab and paclitaxel in negative estrogen receptor participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel (ER-) | Trastuzumab + BKM120 PBO + Paclitaxel (ER-)
Number analyzed (Participants) | 9 | 10
Percentage of participants | 33.3 [7.5 to 70.1] | 60.0 [26.2 to 87.8]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel (ER-) vs Trastuzumab + BKM120 PBO + Paclitaxel (ER-); For ER- participants - pCR; Test type: Superiority; p = 0.949, Fisher Exact; (one-sided)

13. Secondary Outcome: Percentage of Participants With Objective Response Rates by Hormone Receptor Status - Positive Estrogen Receptor (ER+)
Description: Objective response rate = Complete Response + Partial Response rate, measured by US bidimentional ulltrasound (or MRI) and assessed by world health organization (WHO) criteria. CR: Complete disappearance of all tumor signs in the breast as assessed by ultrasound or MRI. The response of the axillary nodes was not to be considered. PR: Reduction in the product of the two largest perpendicular diameters of the primary tumor size by 50% or more assessed by ultrasound or MRI. In patients with multifocal or multicentric disease, the lesion with the largest diameters should be chosen for follow-up. The response of the axillary nodes was not to be considered.
Time Frame: After Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Trastuzumab + BKM120 + Paclitaxel (ER+): BKM120 (oral, pan-class I PI3K inhibitor) in combination with trastuzumab and paclitaxel in positive estrogen receptor participants.
- Trastuzumab + BKM120 PBO + Paclitaxel (ER+): BKM120 placebo in combination with trastuzumab and paclitaxel in positive estrogen receptor participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel (ER+) | Trastuzumab + BKM120 PBO + Paclitaxel (ER+)
Number analyzed (Participants) | 16 | 15
Percentage of participants | 68.8 [41.3 to 89.0] | 33.3 [11.8 to 61.6]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel (ER+) vs Trastuzumab + BKM120 PBO + Paclitaxel (ER+); For ER+ participants - ORR; Test type: Superiority; p = 0.053, Fisher Exact; (one-sided)

14. Secondary Outcome: Percentage of Participants With Objective Response Rates by Hormone Receptor Status - Negative Estrogen Receptor (ER-)
Description: as for outcome 13
Time Frame: After Week 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel (ER-) | Trastuzumab + BKM120 PBO + Paclitaxel (ER-)
Number analyzed (Participants) | 9 | 10
Percentage of participants | 33.3 [7.5 to 70.1] | 60.0 [26.2 to 87.8]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel (ER-) vs Trastuzumab + BKM120 PBO + Paclitaxel (ER-); For ER- participants - ORR; Test type: Superiority; p = 0.949, Fisher Exact; (one-sided)

15. Secondary Outcome: Percentage of Participants With Remaining Ductal Carcinoma in Situ (DCIS) (ypTis)
Description: This included participants at definitive surgery irrespective of lymph node status
Time Frame: 18 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 12.0 [2.5 to 31.2] | 12.0 [2.5 to 31.2]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; Test type: Superiority; p = 0.666, Fisher Exact; (one-sided)

16. Secondary Outcome: Percentage of Participants With Node-negative Disease at Definitive Surgery (ypN0)
Description: Node-negative disease at definitive surgery (ypN0) were considered as binary variables of 'response' versus 'non response'.
Time Frame: 18 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
Number analyzed (Participants) | 25 | 25
Percentage of participants | 52.0 [31.3 to 72.2] | 60.0 [38.7 to 78.9]
Statistical Analysis 1: Comparison: Trastuzumab + BKM120 + Paclitaxel vs Trastuzumab + BKM120 PBO + Paclitaxel; Test type: Superiority; p = 0.803, Fisher Exact; (one-sided)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for a median of approximately 18 months. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of approx. 18 months.
Description: All cause mortality (deaths) was collected for as long as participants could be contacted from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to a maximum of approx. 18 months.
Arm/Group | Trastuzumab + BKM120 + Paclitaxel | Trastuzumab + BKM120 PBO + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 8/25 | 2/25
Other Adverse Events (participants affected / at risk) | 21/25 | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + BKM120 + Paclitaxel (N=25) | Trastuzumab + BKM120 PBO + Paclitaxel (N=25)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Catheter site pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + BKM120 + Paclitaxel (N=25) | Trastuzumab + BKM120 PBO + Paclitaxel (N=25)
Anemia (Blood and lymphatic system disorders) | 17 | 18
Leukopenia (Blood and lymphatic system disorders) | 11 | 15
Lymphopenia (Blood and lymphatic system disorders) | 11 | 8
Neutropenia (Blood and lymphatic system disorders) | 6 | 9
Thrombopenia (Blood and lymphatic system disorders) | 4 | 0
Cardiac disorders not yet listed (Cardiac disorders) | 1 | 3
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 2
Eye disorders (Eye disorders) | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhea (Gastrointestinal disorders) | 15 | 10
Dysgeusia (Gastrointestinal disorders) | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Mucositis (Gastrointestinal disorders) | 19 | 12
Nausea (Gastrointestinal disorders) | 11 | 8
Other gastrointestinal disorders (Gastrointestinal disorders) | 7 | 7
Upper abdominal pain (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2
Chills (General disorders) | 1 | 4
Fatigue (General disorders) | 13 | 14
Oedema (General disorders) | 3 | 8
Other general disorders and administration site conditions (General disorders) | 2 | 1
Allergic reactions (Immune system disorders) | 3 | 1
Fever without neutropenia (Infections and infestations) | 7 | 3
Infection (Infections and infestations) | 12 | 19
Injury and poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 2
Decreased calcium (Investigations) | 9 | 11
Decreased potassium (Investigations) | 6 | 2
Decreased serum albumin (Investigations) | 5 | 2
Decreased sodium (Investigations) | 9 | 7
Increased ALT (Investigations) | 21 | 18
Increased AP (Investigations) | 6 | 6
Increased AST (Investigations) | 19 | 9
Increased FPG (Investigations) | 13 | 8
Increased GGT (Investigations) | 8 | 7
Increased aPTT (Investigations) | 5 | 6
Increased potassium (Investigations) | 3 | 11
Increased serum creatinine (Investigations) | 1 | 2
Increased sodium (Investigations) | 4 | 2
Increased total bilirubin (Investigations) | 2 | 0
Increased total cholesterol (Investigations) | 14 | 14
Increased triglycerides (Investigations) | 5 | 6
Increased uric acid (Investigations) | 6 | 10
Anorexia (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Other musculo-skeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 9 | 4
Headache (Nervous system disorders) | 2 | 8
Other neurological disorder (Nervous system disorders) | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 16
Anxiety (Psychiatric disorders) | 5 | 3
Depression (Psychiatric disorders) | 6 | 8
Insomnia (Psychiatric disorders) | 3 | 4
Psychiatric disorders (Psychiatric disorders) | 2 | 0
Renal and urinary disorders (Renal and urinary disorders) | 2 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Other respiratory and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 5 | 5
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 | 12
Rash other than macular-papular or NOS (Skin and subcutaneous tissue disorders) | 8 | 8
Hot flushes (Vascular disorders) | 5 | 7
Vascular disorders (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.